CLINICAL TRIAL: NCT00715663
Title: A Multi-center, Prospective, Non-interventional Evaluation of Efficacy, Safety and Convenience of Using NovoMix® 30 FlexPen® as Monotherapy, or in Combination With OHA, in Treatment of Type 2 Diabetic Patients in Routine Clinical Practice: A Post-Marketing Surveillance Study
Brief Title: Observational Study to Evaluate Safety, Efficacy and Convenience of Using NovoMix® 30 FlexPen® in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NOPEN3-1891
Record Dates: First submitted 2008-07-14; First posted 2008-07-15 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Delivery Systems
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — No intervention is done. For study drug, start dose and frequency of administration to be prescribed by the physician as a result of normal clinical evaluation
  Other Names: NovoMix® 30

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to evaluate safety, efficacy and convenience in using NovoMix® 30 FlexPen® in type 2 diabetes under normal clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* All patients with type 2 diabetes, not adequately controlled on their current therapy, who were prescribed NovoMix® 30 FlexPen® as monotherapy, or in combination with OHA, in accordance with the approved labeling, are eligible for the survey.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with type 2 diabetes, inadequately controlled on their current therapy, who are prescribed NovoMix® 30 FlexPen® as monotherapy, or in combination with OHA, in accordance with the approved labelling.
Sampling Method: Non-Probability Sample
Enrollment: 1584 (Actual)
Dates: Start 2007-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | after 12 weeks of therapy
Change in post-prandial glucose (PPG) | after 12 weeks of therapy
Change in fasting plasma glucose (FPG) | after 12 weeks of therapy
Change in prandial glucose increment (PGI) | after 12 weeks of therapy
Incidence of hypoglycaemia and other adverse drug reaction | after 12 weeks of therapy
Patient and doctor's convenience | after 12 weeks of therapy

SECONDARY OUTCOMES:
Response of different patient profiles to NovoMix 30 therapy and patient profiles considered eligible for insulin treatment in physicians' routine clinical practice | For the duration of the study
Patient satisfaction on devices | after 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Jakarta, Indonesia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com